CLINICAL TRIAL: NCT01688102
Title: The Effect of Oral Vitamin D Versus Narrow-Band UV-B Exposure on the Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Manish Ponda, Assistant Professor of Clinical Investigation, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPO-0787
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Ultraviolet Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Vitamin D3 (Active Comparator): Participants will receive oral vitamin D3 50,000 units weekly for 8 weeks. If 25(OH)D levels remain <35 ng/ml, subjects will receive additional doses of oral vitamin D.
  Interventions: Dietary Supplement: Oral Vitamin D3
- Ultraviolet Light (Active Comparator): Subjects will receive 16 treatments with ultraviolet light (narrow band UVB) over 8 weeks. If 25(OH)D levels remain <35 ng/ml, subjects will receive additional doses of narrow band UVB.
  Interventions: Radiation: Ultraviolet Light

INTERVENTIONS:
Dietary Supplement: Oral Vitamin D3 — 50,000 units orally, each week x8 weeks; supplemental doses of 50,000 units orally, each month thereafter as needed
  Arms: Oral Vitamin D3
Radiation: Ultraviolet Light — 16 treatments, 2-3 times weekly over 8 weeks; initial dose 45-75 seconds, whole-body exposure except face and groin, increasing by 10% as tolerated, to a maximum of 4.5 minutes
  Arms: Ultraviolet Light

SUMMARY:
Participants in this study will be randomized to receive either oral vitamin D pills OR ultraviolet light treatment. The investigators will compare how these two methods of raising vitamin D levels will affect cholesterol levels.

DETAILED DESCRIPTION:
Potential subjects will be screened for eligibility, including serum 25(OH)D levels <20ng/ml. Eligible subjects will be randomly assigned to receive either: 1) oral vitamin D3, 50,000 units weekly for 8 weeks or 2) narrow-band UVB radiation, 2 treatments/wk for 8 weeks. Duration of treatment will be based on skin type. After 8 weeks, 25(OH)D levels will be measured monthly. For participants with levels <35 ng/ml, additional doses of oral vitamin D3 or UV radiation will be administered.

A subset of participants from both groups will participate in a skin biopsy cohort, where skin biopsies are obtained before and after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Vitamin D 25-OH level < 20 ng/ml

Exclusion Criteria:

1. Serum calcium > 10.5 mg/dl
2. Serum phosphorus > 5.5 mg/dl
3. Serum parathyroid hormone (PTH) level < 12 pg/ml
4. LDL cholesterol > 190 mg/dl
5. History of recent acute infection (within 1 month)
6. Glomerular filtration rate(GFR) < 60 mL/min
7. Liver Function tests indicative of liver disease (aspartate aminotransferase (AST) or alanine transferase (ALT) > 3x ULN)
8. Current use of Vitamin D > 400 IU/day
9. Current use of any statins, fibrates, niacin, or ezetimibe
10. Current use of any medications affecting sensitivity to UV light
11. Pregnancy (self-reported)
12. Intentional UV exposure (e.g. tanning bed use) in the last 2 weeks or planned use while participating in the study
13. history of malignancy not in remission (> 6 months)
14. History of malignant melanoma
15. Participation in an investigational drug study within 30 days of the screening visit
16. Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.
17. History of any non-melanoma skin cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Ponda, MD MS, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

REFERENCES:
- [Derived] Ponda MP, Liang Y, Kim J, Hutt R, Dowd K, Gilleaudeau P, Sullivan-Whalen MM, Rodrick T, Kim DJ, Barash I, Lowes MA, Breslow JL. A randomized clinical trial in vitamin D-deficient adults comparing replenishment with oral vitamin D3 with narrow-band UV type B light: effects on cholesterol and the transcriptional profiles of skin and blood. Am J Clin Nutr. 2017 May;105(5):1230-1238. doi: 10.3945/ajcn.116.150367. Epub 2017 Feb 22. PMID 28228421

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Started | 60 | 58
Completed | 44 | 40
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Vitamin D3 | Ultraviolet Light | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 39 (12) | 42 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 28 | 25 | 53
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL Cholesterol Level
Time Frame: baseline and 6 months or last observation carried forward (minimum 2 months)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
mg/dl | 3.2 (18.4) | 1.4 (17.8)

2. Secondary Outcome: Change in Total Cholesterol
Description: Change in Total Cholesterol
Time Frame: baseline and 6 months or last observation carried forward (minimum 2 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
mg/dL | 4.1 (22) | 2.0 (18.8)

3. Secondary Outcome: Change in HDL Cholesterol
Time Frame: baseline and 6 months or last observation carried forward (minimum 2 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
mg/dL | 0.2 (8.1) | 0.3 (8.4)

4. Secondary Outcome: Change in Triglycerides
Time Frame: baseline 6 months or last observation carried forward (minimum 2 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
mg/dL | 2.6 (35.4) | 1.7 (42.0)

5. Secondary Outcome: Change in C Reactive Protein
Time Frame: baseline and 6 months
Population: Data analyzed are only for those who completed 6 months of therapy
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 44 | 40
mg/L | 1.88 (6.87) | -.11 (5.1)

6. Secondary Outcome: Change in 25(OH)D
Time Frame: baseline vs. 6 months
Population: Data only for those who completed 6 months of therapy
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 44 | 40
ng/ml | 18.7 (8.0) | 15.6 (8.2)

7. Secondary Outcome: Change in Serum Calcium
Time Frame: baseline vs. 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 44 | 40
mg/dL | .09 (.35) | .07 (.29)

8. Secondary Outcome: Change in Parathyroid Hormone (PTH)
Time Frame: baseline vs.6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 44 | 40
pg/mL | -5 (19) | -9 (31)

9. Other Pre Specified Outcome: Correlation Between Change in LDL Cholesterol and Change in Calcium
Description: The Correlation between change in LDL cholesterol and change in serum calcium
Time Frame: 2 months
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
Pearson correlation coefficient | 0.24 | .16

10. Other Pre Specified Outcome: Correlation Between Change in LDL Cholesterol and Change in PTH
Time Frame: 2 months
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 60 | 58
Pearson correlation coefficient | -.01 | .18

11. Other Pre Specified Outcome: Gene Expression Changes in Peripheral Blood
Description: Interferon response genesets (curated by GSEA). Values are presented as the normalized enrichment score, a metric of gene upregulation (when positive) or down-regulation (when negative), normalized for gene set size. This is a useful basis for comparison for direction and degree of change between treatment groups and GSEA genesets.
Time Frame: baseline vs. 2 months
Measure: Number; unit: GSEA Normalized Enrichment Score
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 15 | 13
GSEA Normalized Enrichment Score
  Interferon-alpha response | 4.14 | -4.05
  Interferon-gamma response | 3.41 | -4.86

12. Other Pre Specified Outcome: Gene Expression Changes in Skin
Description: as for outcome 11
Time Frame: baseline vs. 2 months
Measure: Number; unit: GSEA Normalized Enrichment Score
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Number analyzed (Participants) | 9 | 7
GSEA Normalized Enrichment Score
  Interferon-alpha response | 2.08 | -2.43
  Interferon-gamma response | 2.12 | -2.00

ADVERSE EVENTS:
Arm/Group | Oral Vitamin D3 | Ultraviolet Light
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/58
Other Adverse Events (participants affected / at risk) | 7/60 | 21/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Vitamin D3 (N=60) | Ultraviolet Light (N=58)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Vitamin D3 (N=60) | Ultraviolet Light (N=58)
Skin erythema/burn (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (15)
GI Distress (Gastrointestinal disorders) | 6 (9) | 2 (2)
Skin dryness/irritation (Skin and subcutaneous tissue disorders) | 1 (3) | 8 (9)
Constipation/Hemmorhoids (Gastrointestinal disorders) | 4 (4) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes